CLINICAL TRIAL: NCT00624026
Title: Prospective, Single-arm, Multicenter, Open-label Study to Investigate the Efficacy and Tolerability of the Once Daily (OD) Memantine Treatment
Brief Title: Memantine - Communication Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRZ 90001-0608/1
Record Dates: First submitted 2008-02-14; First posted 2008-02-26 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Memantine-HCl

INTERVENTIONS:
Drug: Memantine-HCl — 20 mg per day (once daily)

SUMMARY:
The study objective is to evaluate the effects of memantine treatment on communication abilities and other cognitive abilities in moderate to severe DAT patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatient at least 50 years of age and at least 8 years of education.
* The patient should have German as a mother-tongue or at least speak the language fluently in order to achieve similar scores in verbal tasks.
* Current diagnosis of probable Alzheimer's disease consistent with NINCDS- ADRDA criteria or with DSM IV TR criteria for Dementia of the Alzheimer's type.
* Mini Mental State Examination (MMSE) total score is less than 20
* Patients treated with any acetylcholinesterase inhibitor (AChEI) may be included, when treatment has started at least 6 months prior screening and was stable during the last 3 months.

Exclusion Criteria:

* Any type of evident aphasia, which may interfere with patient's communication difficulties caused by Alzheimer's disease
* History of severe drug allergy, or hypersensitivity, or patients with known hypersensitivity to amantadine, lactose.
* Evidence (including CT/MRI results) of any clinically significant central nervous system disease other than Alzheimer's disease.
* Modified Hachinski Ischemia score greater than 4 at screening.
* Current evidence of clinically significant systemic disease
* Known or suspected history of alcoholism or drug abuse within the past 10 years.
* Previous treatment with memantine or participation in an investigational study with memantine.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of the memantine OD IR treatment using the Consortium to establish a registry for Alzheimer's Disease (CERAD-NP) total score | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Joerg B. Schulz, MD PhD, Principal Investigator — Center of Neurological Medicine, Goettingen, Germany
Locations (1):
- Central Medical Affairs, Frankfurt am Main, Germany

REFERENCES:
- [Result] Schulz JB, Rainer M, Klunemann HH, Kurz A, Wolf S, Sternberg K, Tennigkeit F. Sustained effects of once-daily memantine treatment on cognition and functional communication skills in patients with moderate to severe Alzheimer's disease: results of a 16-week open-label trial. J Alzheimers Dis. 2011;25(3):463-75. doi: 10.3233/JAD-2011-101929. PMID 21471647